CLINICAL TRIAL: NCT02226224
Title: Endoscopic Ultrasound in Detailed T-staging of Upper GI Malignancies in Vitro
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Yan Yan, Attending physician, Peking University Cancer Hospital & Institute
Other Study IDs: EC1001
Record Dates: First submitted 2014-08-24; First posted 2014-08-27 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Gastrointestinal Neoplasms
Keywords: gastrointestinal neoplasms; endosonography; in vitro; Staging
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- early gastric cancer: EUS examination on the specimen right after surgery mark the deepest invasive site on the specimen
- Locally Advanced Gastric Cancer: EUS examination on the specimen right after surgery mark the deepest invasive site on the specimen
- early esophagus cancer: EUS examination on the specimen right after surgery mark the deepest invasive site on the specimen
- locally advanced esophagus cancer: EUS examination on the specimen right after surgery mark the deepest invasive site on the specimen

SUMMARY:
In our era of personalized treatment, both the prognosis and the choice of therapy for upper GI malignancies depend on the staging before any treatment. Most experts recommend EUS (Endoscopic Ultrasound) as the first line for T-staging but the diagnostic accuracy in clinical practice varies in different centers according to the published data. Neither the discrepancy between EUS and histological findings nor the variation between centers well explained. So the investigators designed this prospective study. In the present study, the investigators performed EUS on the resected specimen after surgery before fixation in formalin, evaluated the invasion of the GI wall, and marked the deepest location with sutures. And try to determine the exact accuracy of EUS staging , find the discrepancy between EUS and histologic findings.

DETAILED DESCRIPTION:
- EUS Examination After the surgery, the specimen is filled with 0.9%NS (normal saline ) without cut open，and put into a container filled with 0.9%NS before fixation in formalin. EUS will be performed on the resected specimen.The endoscopy move from the distal to proximal side along the longitudinal axis of stomach, evaluate the invasion of gastric wall, and mark the deepest point with sutures under the EUS guided. The images were stored .

EUS images the are reviewed by two endoscopists. They are asked to stage the tumor according to the AJCC(American Joint Committee on Cancer) staging system (7th edition) , assign a level of confidence to the staging, and score the quality of the EUS image .

* Histologic Preparations and Examination Carcinoma invasion into each layer of the gastric wall is diagnosed by an experienced pathologist (L.ZW) who is unaware of the findings of the EUS imaging. The marked section will be assessed separately.
* Data analysis The diagnosis between the pathologic findings and EUS prediction will be compared. Whether the marked point was the deepest in pathologic findings is recorded. And the histological section and the EUS image of the marked point is compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients with upper GI carcinoma
* Receive surgery as first treatment

Exclusion Criteria:

* previous surgery involved the upper GI tract

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced upper GI carcinoma receive surgery as first treatment no previous surgery involved the upper GI tract
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2014-06; Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
the consistency between EUS and pathologic determination of tumor depth | 1 month （after careful examination by 2 pathologists）

CONTACTS AND LOCATIONS:
Overall Officials: Yan Yan, Doctor, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China